CLINICAL TRIAL: NCT03973801
Title: Feasibility of Auricular Acupressure as an Adjunct Treatment for Neonatal Abstinence Syndrome (NAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Heather Jackson, Associate in Anesthesiology, Division of Pain Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191023
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Neonatal Abstinence Syndrome; Withdrawal
Keywords: Acupressure
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auricular acupressure (Experimental)
  Interventions: Other: Auricular acupuncture

INTERVENTIONS:
Other: Auricular acupuncture — National Acupuncture Detoxification Association (NADA) protocol for auricular acupressure will be initiated within 24 hours of delivery and continued until withdrawal symptoms measure 6 or less for 12 hours on the modified Finnegan score and/or the morning of expected discharge as in line with standard of care.

SUMMARY:
This study will assess the feasibility of implementing auricular acupressure as an additional non-pharmacologic therapy for neonates at risk for developing neonatal abstinence syndrome (NAS) at Monroe Carrell Jr Children's Hospital at Vanderbilt University Medical Center (VUMC).

DETAILED DESCRIPTION:
NAS is a condition in which newborns experience withdrawal symptoms as a result of in utero exposure to opioids and/or other substances ingested by the mother. The condition has significantly risen over the past 20 years. First line treatments for NAS involve the maximization of non-pharmacologic therapies. NAS management focuses on reducing or eliminating the need for medication management to prevent further developmental complications, promote maternal bonding, and reduce hospital length of stay.

Auricular acupuncture has been used for the treatment of addiction and has demonstrated efficacy in the adult population. Current evidence suggests that acupuncture is safe and beneficial for multiple conditions that impact neonatal and pediatric populations including NAS. Acupressure is a less invasive therapy and may serve as an additional non-pharmacological adjunct to ease the severe discomfort of withdrawal in neonates at risk for NAS.

This study will assess the feasibility of implementing auricular acupressure as an additional non-pharmacologic therapy for neonates at risk for developing neonatal abstinence syndrome (NAS) at Monroe Carrell Jr Children's Hospital at Vanderbilt University Medical Center (VUMC).

ELIGIBILITY:
Inclusion Criteria:

* 37 weeks gestational age or greater
* Maternal age 16 or older
* Substance exposure in utero including opioids, illicit drugs, or other medications that cause neonatal withdrawal

Exclusion Criteria:

* Birth trauma
* Neonatal asphyxia
* Maternal or neonatal infection
* Congenital abnormalities
* Requiring Neonatal Intensive Care Unit (NICU) care

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Percent of eligible patients enrolled | end of study enrollment (about 12 weeks)
Percent of patients prematurely terminating treatment | hospital discharge (about 48-72 hours after delivery)
Percent of participants completing all study assessments | hospital discharge (about 48-72 hours after delivery)
Percent of data collection procedures completed | hospital discharge (about 48-72 hours after delivery)
Percent of missing medical record data | hospital discharge (about 48-72 hours after delivery)

SECONDARY OUTCOMES:
Percent of providers enrolled in 3 day training course for NADA protocol | Prior to start of study enrollment (May 31, 2019)
Percent of providers completing 3 day training course for NADA protocol | Day 3 of training
  Percent of providers completing 3 day training course for NADA protocol: The training course includes a national, standardized curriculum, clinical demonstration and skills lab. Providers are trained in application of acupuncture needles which are placed at the same location as acupressure stickers.
Percent of providers completing clinical competency with NADA protocol | Prior to start of study enrollment (May 31, 2019)
  Percent of providers completing clinical competency with NADA protocol: Following the training course providers must submit pictures to the NADA instructor with a clinical log of 40 appropriately placed acupuncture needles in accordance with the NADA protocol. Training includes
Percent of providers receiving NADA certification | Prior to start of study enrollment (May 31, 2019)
  Percent of providers receiving NADA certification: Once clinical practice is complete and verified by a NADA trainer, providers will receive a NADA certification
Percent of providers receiving credentialing | Prior to start of study enrollment (May 31, 2019)
  Following certification of the providers, competency of acupressure placement on neonates for the specific study protocol will be demonstrated via simulation lab. Providers must perform the acupressure, in accordance with the NADA protocol, on a neonatal manikin, and documentation of the appropriate technique will be completed for credentialing purposes. Providers will submit the NADA certificate, a skills checklist that documents appropriate NADA technique on a neonate manikin, and a neonatal simulation lab certificate for credentialing to perform NADA protocol at VUMC.
Client Satisfaction Questionnaire (CSQ*) Score | Day of discharge (about 48-72 hours after delivery)
  On day of discharge, the parent(s) will receive the Client Satisfaction Questionnaire (CSQ8) to assess parental satisfaction of acupuncture as an additional therapy. The CSQ8 is an 8 item measure of client satisfaction with services. Items are questions inquiring about respondents' opinions and conclusions about services they have received. Response options differ from item to item, but all are based on a four-point scale. The overall score is produced by summing all item responses. CSQ-8 version scores range from 8 to 32, with higher values indicating higher satisfaction.
Intervention Appropriateness Measure (IAM) Score | Day of hospital discharge of baby (about 48-72 hours after delivery)
  Provider and staff acceptability of acupressure as an additional non-pharmacologic treatment will be measured with the Intervention Appropriateness Measure (IAM). The IAM is a four-item measure of the appropriateness of an intervention. Each item of the score is rated on a five point scale where 1 equals completely disagree and 5 equals completely agree. The total score ranges from 5 to 20, with a higher score indicating a higher level of appropriateness.
Acceptability of Intervention Measure (AIM) | Day of hospital discharge of baby (about 48-72 hours after delivery)
  Provider and staff acceptability of acupressure as an additional non-pharmacologic treatment will be measured with the Acceptability of Intervention Measure (AIM). The AIM is a four-item measure of the acceptability of an intervention. Each item of the score is rated on a five point scale where 1 equals completely disagree and 5 equals completely agree. The total score ranges from 5 to 20, with a higher score indicating a higher level of acceptability.
Feasibility of Intervention Measure (FIM) | Day of hospital discharge of baby (about 48-72 hours after delivery)
  Provider and staff acceptability of acupressure as an additional non-pharmacologic treatment will be measured with the Feasibility of Intervention Measure (FIM). The FIM is a four-item measure of the feasibility of an intervention. Each item of the score is rated on a five point scale where 1 equals completely disagree and 5 equals completely agree. The total score ranges from 5 to 20, with a higher score indicating a higher level of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jackson, MSN, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No